CLINICAL TRIAL: NCT02106182
Title: A Multi-center, Prospective, Open-label, Single-arm, 12-weeks, Phase IV Trial to Evaluate the Efficacy and Safety of Silodosin on Nocturia for Patients With Benign Prostatic Hyperplasia
Brief Title: Efficacy and Safety of Silodosin on Nocturia for Patients With Benign Prostatic Hyperplasia
Acronym: BPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JW-SDS-406
Record Dates: First submitted 2014-03-31; First posted 2014-04-08 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Nocturia; Benign Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia; Nocturia; Silodosin; Thrupas
MeSH Terms: conditions — Nocturia; Prostatic Hyperplasia | interventions — silodosin; Clinical Laboratory Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Silodosin (Experimental): Silodosin, 8 mg, once daily, orally administered with dinner for 12 weeks
  Interventions: Drug: Silodosin; Other: Laboratory tests; Other: 3-days voiding diary; Other: 12 weeks

INTERVENTIONS:
Drug: Silodosin
  Other Names: Thrupas Cap
Other: Laboratory tests — Subject's overall health state will be evaluated by clinical laboratory tests.
  Serum chemistry test: Creatinine, Blood Urea Nitrogen(BUN), Aspartate aminotransferase(AST), Alanine aminotransferase(ALT) Urinalysis: Urine Specific Gravity, Urine pH, Urine Protein, Urine Glucose, Urine Ketone, Urine Bilirubin, Urine Urobilinogen, Urine Nitrite, Urine Occult Blood(OB), Urine Red Blood Cell(RBC), Urine White Blood Cell(WBC) Immunoassay: Prostate Specific Antigen(PSA)
Other: 3-days voiding diary — 3-day voiding diaries will be distributed on Visits 1, 2 and 3. Subjects will record incidence of nocturia during 3 days on the diaries within 7 days of Visits 2 (baseline), 3 and 4. The average will be used to confirm the change in incidence of nocturia (at baseline, results from within 1 week from screening may be used but will be excluded for subjects needing wash-out period).
Other: 12 weeks

SUMMARY:
The objective of this study is to determine safety and efficacy of silodosin, which is a treatment for benign prostatic hyperplasia with high selectivity to α1A-receptor, on patients with benign prostatic hyperplasia accompanied by nocturia.

DETAILED DESCRIPTION:
This study is designed as a multi-center, prospective, open-label and single-arm study. Subjects who are willing to provide written informed consent will be enrolled after screening for eligibility criteria. The subjects will be administered with investigational product for 12 weeks and visit as outpatients for evaluation of safety and efficacy at baseline (visit 2) and 4 weeks (visit 3) and 12 weeks (visit 4) after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Males of at least 50 years of age, with current diagnosis of benign prostatic hyperplasia
* Symptoms of nocturia evidenced by ≥2 episodes per night in average according to 3-day voiding diary
* More than total of 8 points on IPSS and 3 points on QoL
* Able to provide written informed consent and to comply with all study procedures

Exclusion Criteria:

* PSA level > 10 ng/㎖ (except patients who had 4 ng/㎖ < PSA level ≤ 10 ng/㎖ 6 months prior to screening and identified as negative from biopsy)
* Symptoms of postural hypotension
* Severe renal disorders or creatinine clearance ≥ 2.0 mg/dL
* Severe hepatic disorders or AST or ALT ≥ 3 x upper limit of normal (ULN)
* Severe cardiac disorders or development or diagnosis of vascular disorder (unstable angina, myocardial infarction, cerebral infarction, cerebral hemorrhage, coronary artery bypass graft, etc) 6 months prior to enrollment
* Any disorder of the gastrointestinal system which could result in altered digestion or absorption, history of gastrointestinal tract surgery except ecphyadectomy
* Patients with bladder cancer, cystolith or urethral stricture
* Patients with neurogenic bladder
* History of acute urinary retention
* Indwelling catheter or self intermittent catheterization
* Patients with pyuria 1 month prior to screening
* History of prostatic cancer
* History of prostatic surgery
* Patients with uncontrolled chronic disease
* Alcoholism or sustained drug dependent abuse 1 year prior to screening
* Hypersensitivity to α1A-receptor blockers
* Administration of following drugs within according periods prior to screening - 2 weeks: Antimuscarinic agents (Tolterodine, Trospium, Solifenacin, Fesoterodine, Propiverine, Oxybutynin, Flavoxate, etc), Anticholinesterase agents (Neostigmine methylsulfate, etc), Cholinergic agonists (Bethanechol Cl, etc), Benign prostatic hyperplasia agents (Tamsulosin HCl, Prazosin HCl, Terazosin HCl, Doxazosin mesylate, Silodosin, Naftopidil, etc), Tricyclic antidepressants (Amitriptyline, Clomipramine, Dosulepin, Doxepin, Imipramine, Quinupramine, etc), 6 months: 5-α-Reductase Inhibitors (Finasteride, Dutasteride)
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2016-03-02 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of nocturia | 12 weeks
  Descriptive statistics for incidence of nocturia will be provided for each visit. Paired t-test or Wilcoxon's signed rank test will be used for assessment of change from baseline to after 12 weeks of treatment.

SECONDARY OUTCOMES:
Mean change in International Prostate Symptom Score(IPSS) from baseline | 12 weeks
  Descriptive statistics for secondary efficacy outcome measures will be provided for each visit. Assessment will be performed on whether the change from baseline to after 12 weeks of treatment has difference. For successive data, paired t-test or Wilcoxon's signed rank test will be used for assessment of change from baseline to after 12 weeks of treatment.
Mean change in Quality of Life(QoL) scores from baseline | 12 weeks
  Descriptive statistics for secondary efficacy outcome measures will be provided for each visit. Assessment will be performed on whether the change from baseline to after 12 weeks of treatment has difference. For successive data, paired t-test or Wilcoxon's signed rank test will be used for assessment of change from baseline to after 12 weeks of treatment.
Mean change in Overactive Bladder Symptom Score(OABSS) from baseline | 12 weeks
  Descriptive statistics for secondary efficacy outcome measures will be provided for each visit. Assessment will be performed on whether the change from baseline to after 12 weeks of treatment has difference. For successive data, paired t-test or Wilcoxon's signed rank test will be used for assessment of change from baseline to after 12 weeks of treatment.
Mean change in International Consultation on Incontinence modular Questionnaire-Nocturia(ICIQ-N) from baseline | 12 weeks
  Descriptive statistics for secondary efficacy outcome measures will be provided for each visit. Assessment will be performed on whether the change from baseline to after 12 weeks of treatment has difference. For successive data, paired t-test or Wilcoxon's signed rank test will be used for assessment of change from baseline to after 12 weeks of treatment.
Mean change in Questions 3, 5 and 6 (voiding symptoms) of IPSS from baseline | 12 weeks
  Descriptive statistics for secondary efficacy outcome measures will be provided for each visit. Assessment will be performed on whether the change from baseline to after 12 weeks of treatment has difference. For successive data, paired t-test or Wilcoxon's signed rank test will be used for assessment of change from baseline to after 12 weeks of treatment.
Mean change in Question 1 (postvoiding symptoms) of IPSS from baseline | 12 weeks
  Descriptive statistics for secondary efficacy outcome measures will be provided for each visit. Assessment will be performed on whether the change from baseline to after 12 weeks of treatment has difference. For successive data, paired t-test or Wilcoxon's signed rank test will be used for assessment of change from baseline to after 12 weeks of treatment.
Mean change in Questions 2, 4 and 7 (storage symptoms) from baseline | 12 weeks
  Descriptive statistics for secondary efficacy outcome measures will be provided for each visit. Assessment will be performed on whether the change from baseline to after 12 weeks of treatment has difference. For successive data, paired t-test or Wilcoxon's signed rank test will be used for assessment of change from baseline to after 12 weeks of treatment.
Ratio of subjects with ≥ 25% decrease in incidence of nocturia | 12 weeks
Ratio of subjects with ≥ 25% decrease in IPSS | 12 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Bucheon St.Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Pusan Natonal University Hospital, Busan
  - Eulji University Hospital, Daejeon
  - Hanyang University Hospital, Seoul
  - Soon Chun Hyang University Hospital, Seoul